CLINICAL TRIAL: NCT02213848
Title: Effect of Calcium Chloride on Recovery From Neuromuscular Blockade in Patients Undergoing General Anesthesia
Brief Title: Effect of Calcium Chloride on Recovery From Neuromuscular Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Deok Man Hong, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Calcium RNMB
Record Dates: First submitted 2014-08-04; First posted 2014-08-12 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2014-08

CONDITIONS: Residual Neuromuscular Blockade
Keywords: Neuromuscular blockade reversal; TOF ratio; Calcium chloride
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium (Experimental): Administration of calcium chloride 5 mg/kg along with neostigmine 25 mcg/kg + atropine 15 mcg/kg
  Interventions: Drug: Calcium
- control (Placebo Comparator): In the control group, all the procedures were the same with calcium group, except for the fact that calcium chloride is not administered
  Interventions: Drug: control

INTERVENTIONS:
Drug: Calcium — Administration of calcium chloride 5 mg/kg along with neostigmine 25 mcg/kg + atropine 15 mcg/kg
  Arms: Calcium
Drug: control — In the control group, all the procedures were the same with calcium group, except for the fact that calcium chloride is not administered
  Arms: control

SUMMARY:
The purpose of this study is to evaluate the effect of calcium chloride against residual neuromuscular blockade at the end of general anesthesia

DETAILED DESCRIPTION:
During general anesthesia, neuromuscular blocking agent is administered to facilitate endotracheal intubation and the view of operative field. The neuromuscular blockade should be reversed at the end of anesthesia to recover spontaneous breathing of the patient.

Residual neuromuscular blockade (RNMB) is defined as train of-four ratio < 0.9. RNMB is a risk factor for postoperative pulmonary complication and increases postoperative mortality. Neostigmine is acetylcholinesterase inhibitor routinely used at the end of anesthesia to prevent RNMB. A meta-analysis, however, showed that 40 percent of patients who received intermediate-acting neuromuscular blocking agent during anesthesia showed RNMB in PACU.

Calcium triggers the release of acetylcholine from the motor nerve terminal and enhances excitation-contraction coupling in muscle. Increasing calcium concentrations decreased the sensitivity to dTc and pancuronium in an animal muscle-nerve model. The effect of calcium chloride on residual neuromuscular blockade is not studied yet.

The purpose of this study is to evaluate the effect of calcium chloride on residual neuromuscular blockade at the end of general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yr
* Body mass index 15.0-25.0 kg/m2
* American Society of Anesthesiologists physical status I-III
* Scheduled for elective surgery with an expected duration of more than 60 min under general anesthesia with endotracheal intubation

Exclusion Criteria:

* Suspected difficulty airway
* Bronchial asthma, chronic obstructive pulmonary disease
* Neuromuscular disease
* Hepatic or renal dysfunction.
* Taking medications that might influence the effect of neuromuscular blocking agents
* Allergy to the medication that used in this trial
* Pregnant, or breastfeeding state
* Suspected malignant hyperthermia
* Contraindication to the medication that used in this trial
* Hypercalcemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Time to train of-four ratio of 0.9. | At 10 minutes (expected aeverage) after the surgery
  Train of-four will be measured using acceleromyograph.

SECONDARY OUTCOMES:
Train of-four ratio | At 5, 10, 20 minutes after the administration of reversal drug
  Train of-four will be measured using accelerography.
Length of PACU stay | At 60 minutes (expected average) after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Chang Kim, M.D., Ph. D., Study Director — Seoul National University Hospital; Jae Woo Ju, M.D., Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea